CLINICAL TRIAL: NCT02836392
Title: CRQ Survey Study: Clinical Research Questionnaire of Oncology Patients - A Nationwide Survey
Status: Completed | Type: Observational
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Other Study IDs: ICORG 15-43
Record Dates: First submitted 2016-06-27; First posted 2016-07-19 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Questionnaire

SUMMARY:
This is a translational, multicentre questionnaire study. The study design follows that of a cross sectional, quantitative research approach. Data collection will involve self-administered, paper-based questionnaires. The method of data collection allows for a large sample size without major expense. The questionnaires are comprised of several questions examining areas such as demographic details, cancer diagnosis, understanding of the term 'clinical trials', attitudes to personal participation in cancer clinical research and the experience of patients who previously participated in a cancer clinical trial. The study will be opened in all interested hospitals in Ireland following initiation of the study at each site. Questionnaire completion will be seen as implied informed consent and no formal consent will need to be signed by the patient. The paper-based questionnaire responses will be electronically and anonymously recorded in a computer database to facilitate analysis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of malignancy
* Aged 18 years or older
* Ability to complete the questionnaire or independently or with the help of a friend, relative, or staff member of the oncology department

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a translational, multicentre questionnaire study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Oncology patients' understanding of the term 'clinical trials' and their attitudes towards personal participation in cancer clinical research will be evaluated by questionnaire. | 1 year

SECONDARY OUTCOMES:
The patient related factors, including level of education and socioeconomic status that influence their decision regarding participation in a cancer clinical trial (CCT) will be explored by questionnaire. | 1 year
The patients' experience surrounding the discussion regarding CCT participation and their actual experience when enrolled in a CCT will be investigated by questionnaire. | 1 year

CONTACTS AND LOCATIONS:
Locations (14):
- Ireland (14):
  - University Hospital Waterford, Waterford, Co Waterford
  - AMNCH, Tallaght, Dublin 24
  - St Vincent's University Hospital, Elm Park, Dublin 4
  - Beaumont Hospital, Beaumont Road, Dublin
  - Bon Secours Hospital, Cork
  - Cork University Hospital, Cork
  - Saint Luke's Hospital Rathgar, Dublin
  - Beacon Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St James Hospital, Dublin
  - University Hospital Galway, Galway
  - Letterkenny General Hospital, Letterkenny
  - University Hospital Limerick, Limerick
  - Sligo University Hospital, Sligo

IPD SHARING:
Plan to Share IPD: Yes